CLINICAL TRIAL: NCT00762918
Title: Vitamin D and Its Non-Classic Roles in Cystic Fibrosis
Brief Title: Vitamin D3 for the Treatment of Low Vitamin D in Cystic Fibrosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Andrea Kelly, The Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-12-5688
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Cystic Fibrosis; Vitamin D Deficiency
Keywords: cystic fibrosis; vitamin d; inflammation
MeSH Terms: conditions — Cystic Fibrosis; Vitamin D Deficiency; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: cholecalciferol — cholecalciferol 5000 IU capsule by mouth daily for 3 months
  Other Names: Vitamin D3

SUMMARY:
Vitamin D deficiency is common in cystic fibrosis. Vitamin D deficiency frequently persists despite aggressive treatment with ergocalciferol, a vitamin D preparation also known as vitamin D2. Cholecalciferol, a vitamin D preparation also known as vitamin D3,may work better to increase vitamin D levels.

Vitamin D is important for absorption of calcium from the diet and bone health. Vitamin D more recently has been found to play a role in regulating the normal inflammatory process. Since cystic fibrosis is a state of excessive inflammation, vitamin D may be playing a role in cystic fibrosis.

We hypothesize: cholecalciferol will work better to increase vitamin D levels in patients iwth cystic fibrosis and that it will have an effect on markers of inflammation.

DETAILED DESCRIPTION:
Vitamin D deficiency is common in cystic fibrosis (CF) and persists despite relatively high doses of ergocalciferol, vitamin D2. Replacement has traditionally been focused upon maintenance of calcium and phosphorus homeostasis and bone health. However, non-classic roles of vitamin D have become increasingly recognized and the contribution of vitamin D deficiency to non-bone disorders has become apparent. Vitamin D deficiency has been associated with increased risk of a variety of cancers, autoimmune diseases such as Type 1 diabetes and multiple sclerosis, Type 2 diabetes, tuberculosis, and myopathy. The connection between vitamin D and these disease states likely reflects vitamin D's role as a transcriptional regulator: it participates in cell cycle regulation and in the innate immune system mediates cathelicidin production following activation of toll-like receptors.One hallmark of CF is pulmonary hyper-inflammation with recurrent infections. Additionally, malnutrition and decreased lean muscle mass threaten pulmonary function in CF. While vitamin D and its relation to bone has been explored in CF, the role of vitamin D in inflammation, lean body mass and strength, and pulmonary muscle strength has not been investigated. Moreover, vitamin D replacement has traditionally been with ergocalciferol, vitamin D2. Vitamin D3, cholecalciferol, has a longer half-life and is considered more potent. Thus, cholecalciferol treatment of children and young adults with CF and vitamin D deficiency may be useful for attaining normal vitamin D status and for exploring the impact of vitamin D upon lean body mass, pulmonary muscle strength, and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 10-25 years
2. cystic fibrosis
3. 25-(OH)-D < 20 ng/mL
4. FEV1 > 40% -

Exclusion Criteria:

1. inability to perform pulmonary function or hand-grip tests
2. liver disease (including cirrhosis and portal hypertension) or baseline liver enzymes 21/2-fold greater than the upper limit of normal
3. acute use of glucocorticoids at time of testing
4. acute pulmonary exacerbation at time of testing
5. known non-adherence to enzyme replacement
6. hypercalcemia
7. engages in "suntanning

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
serum 25-hydroxy vitamin D levels | 3 months

SECONDARY OUTCOMES:
body composition | 3 months
inflammatory markers | 3 months
muscles strength | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kelly, MD, Principal Investigator — Children's Hospital of Philadelphia